CLINICAL TRIAL: NCT05288335
Title: Muti-center Clinical Trial to Evaluate the Safety and Efficacy of Two Types of Circular Column Modulated Lenses for Delaying the Progression of Myopia
Brief Title: Evaluate the Safety and Efficacy of Two Types of Circular Column Modulated Lenses for Delaying the Progression of Myopia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TianjinEH-myopia progression
Record Dates: First submitted 2022-02-10; First posted 2022-03-21 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Circular cylindrical mirror modulated frame glasses (compact) (Experimental): Subjects that were randomized to receive the Circular cylindrical mirror modulated frame glasses (compact) throughout the entire course of the study.
  Interventions: Device: Circular cylindrical mirror modulated frame glasses (compact)
- Circular cylindrical mirror modulated frame glasses (strong defocus) (Experimental): Subjects that were randomized to receive the Circular cylindrical mirror modulated frame glasses (strong defocus) throughout the entire course of the study.
  Interventions: Device: Circular cylindrical mirror modulated frame glasses (strong defocus)
- single vision frame glasses (Experimental): Subjects that were randomized to receive the single vision frame glasses throughout the entire course of the study.
  Interventions: Device: single vision frame glasses

INTERVENTIONS:
Device: Circular cylindrical mirror modulated frame glasses (compact) — Circular cylindrical mirror modulated frame glasses (compact)
  Arms: Circular cylindrical mirror modulated frame glasses (compact)
Device: Circular cylindrical mirror modulated frame glasses (strong defocus) — Circular cylindrical mirror modulated frame glasses (strong defocus)
  Arms: Circular cylindrical mirror modulated frame glasses (strong defocus)
Device: single vision frame glasses — single vision frame glasses
  Arms: single vision frame glasses

SUMMARY:
Clinical trial to evaluate the safety and effectiveness of two kinds of ring band cylindrical lens in delaying the progression of myopia

DETAILED DESCRIPTION:
Two-hundered and forty children aged 6-13 will be recruited and allocated to three groups. Subjects that were randomized to receive Circular cylindrical mirror modulated frame glasses (compact), Circular cylindrical mirror modulated frame glasses (strong defocus) or single vision frame glasses, respectively.

Primary outcome measure ocular axial length and the secondary indicator is spherical equivalent after cycloplegia.

ELIGIBILITY:
Inclusion Criteria:

1. 6-13 years old;
2. SER: -0.75 to -5.00 dioptres (D). Astigmatism and anisometropia of 1.50 D or less;
3. Monocular best corrected visual acuity (VA) of 1.0 or better;
4. Acceptance of random group allocation and the masked study design
5. Voluntarily participate in the clinical trial and sign the informed consent;

Exclusion Criteria:

1. Strabismus.
2. Ocular and systemic abnormalities.
3. Prior experience of myopia control.
4. Only one eye meets the inclusion criteria.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-10-15 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in ocular axial length in a year | baseline, 12 months
  The ocular axial length was measured by AL-scan

SECONDARY OUTCOMES:
Changes in cycloplegic objective spherical equivalent in a year | baseline, 12 months
  The cycloplegic objective spherical equivalent was evaluated by a autorefractor

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoqin Chen, MD, Principal Investigator — Tianjin Eye Hospital
Locations (1):
- Tianjin Eye Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bao J, Yang A, Huang Y, Li X, Pan Y, Ding C, Lim EW, Zheng J, Spiegel DP, Drobe B, Lu F, Chen H. One-year myopia control efficacy of spectacle lenses with aspherical lenslets. Br J Ophthalmol. 2022 Aug;106(8):1171-1176. doi: 10.1136/bjophthalmol-2020-318367. Epub 2021 Apr 2. PMID 33811039
- [Derived] Muller J, Chen X, Ohlendorf A, Li L, Wahl S. Method comparison and overview of refractive measurements in children: implications for myopia management. BMJ Open Ophthalmol. 2024 Mar 1;9(1):e001322. doi: 10.1136/bmjophth-2023-001322. PMID 38429067